CLINICAL TRIAL: NCT00389454
Title: Acetaminophen Concentration in Cerebrospinal Fluid in Infants
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 93/03
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2006-08

CONDITIONS: Fever
Keywords: Acetaminophen; Fever; cerebro spinal fluid; Infants
MeSH Terms: conditions — Fever

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Acetaminophen is the most commonly used drug in children. Inhibition of COX-3 in the brain has been suggested as the primary central mechanism by which acetaminophen decrease pain and possibly fever. However there is very limited data about acetaminophen concentrations in the brain and no such data is available for newborns. The objective of the current study is to describe concentrations of acetaminophen in the fluid around the brain of infants after administration of acetaminophen.

DETAILED DESCRIPTION:
The mechanism by which acetaminophen causes analgesia and antipyretic effect is not entirely clear. Recently a new COX isoenzyme was identified and termed COX 3. In humans this isoenzyme is most abundant in cerebral cortex and heart. Inhibition of COX-3 could represent a primary central mechanism by which acetaminophen decrease pain and possibly fever (10). An effect on of acetaminophen on presynaptic 5-HT(2) receptors in the hypocampus has been demonstrated (11) suggesting again that the primary effect of acetaminophen is in the CNS.

Many studies (12-16) described the pharmacokinetics of oral and rectal acetaminophen in infants and neonates. Yet, the data on acetaminophen concentrations in the CSF is very limited. Two studies in adults (17;18) used intravenous propacetamol and described concentrations of acetaminophen in the plasma and CSF. Acetaminophen was detected as early as 15 minutes after the administration and reached peak concentrations in the CSF at the 4th hour. A small study (19) of nine children who had indwelling ventricular drains found that cerebrospinal fluid concentrations lagged behind those of plasma with an equilibration half time of 0.72 h. This study did not describe CSF concentrations in neonates and used a dose of 40mg/kg, which is higher than the recommended dose in children. To the best of our knowledge there is no data on acetaminophen CSF concentrations in neonates.

The objective of the current study is to describe concentrations of acetaminophen in the CSF of infants after single administration of acetaminophen. A better understanding of the pharmacokinetics of acetaminophen and its penetration into the CSF will enable us to better predict the effects of this commonly used drug.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1week - 2 years
* Rectal temperature > 38.0OC
* A sepsis work up is indicated
* Acetaminophen was given prior to lumbar puncture (LP)

Exclusion Criteria:

* Hypersensitivity to acetaminophen
* Known metabolic disorder
* Known liver or kidney disease
* Hydrocephalus
* Informed consent could not be obtained from a legal guardian

Ages: 1 Week to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-01; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eran Kozer, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Pediatric Emergency Unit Assaf Harofeh Medical center, Ẕerifin, Israel